CLINICAL TRIAL: NCT00159640
Title: A Multi-Center, Randomized, Double Blind, Dose-Response, Placebo And Gabapentin Controlled Study Of PD-217,014 In The Treatment Of Postherpetic Neuralgia
Brief Title: Placebo Controlled Dose-Response Study Of PD-217,014 In The Treatment Of Postherpetic Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4451006
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: PD-217,014

SUMMARY:
The purpose of this study is to determine the effectiveness of PD-217,014 in the treatment of chronic pain following a shingles infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after the healing of shingles skin rash.
* Patients at screening must have a score >=40 mm on the pain visual analogue scale.

Exclusion Criteria:

* Patients with poor renal function.
* Patients with other severe pain, that may impair the self-assessment of the pain due to shingles.
* Patients with abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315
Dates: Start 2004-02

PRIMARY OUTCOMES:
To characterise the effectiveness of PD-217,014 in the treatment of chronic pain. A numerical pain intensity rating scale is used to assess pain and a mean endpoint (week 4) pain score change from baseline is calculated.

SECONDARY OUTCOMES:
- Assess the effect of PD-217,014 on responder rate based on the primary endpoint, mean endpoint sleep interference score and the SF-McGill questionnaire (change from baseline to week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Australia (7):
  - Pfizer Investigational Site, Warrawong, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Kippa-Ring, Queensland
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Perth, Western Australia
  - Pfizer Investigational Site, Woodville
- Canada (5):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
- Czechia (5):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, CZ-Praha 8
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
- Netherlands (6):
  - Pfizer Investigational Site, Arnhem
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Kampen
  - Pfizer Investigational Site, Roosendaal
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Stadskanaal
- Spain (5):
  - Pfizer Investigational Site, Granada, Granada
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, MALAGA
  - Pfizer Investigational Site, Seville, SEVILLA
  - Pfizer Investigational Site, Barcelona
- United Kingdom (3):
  - Pfizer Investigational Site, Portsmouth, Hants
  - Pfizer Investigational Site, Northampton, Northants
  - Pfizer Investigational Site, London
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4451006&StudyName=Placebo+Controlled+Dose%2DResponse+Study+Of+PD%2D217%2C014+In+The+Treatment+Of+Postherpetic+Neuralgia